CLINICAL TRIAL: NCT05949294
Title: A Phase 1 Dose Escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of ARO-SOD1 in Adult Patients With Amyotrophic Lateral Sclerosis Harboring a Superoxide Dismutase-1 Mutation Considered to be Causative of Amyotrophic Lateral Sclerosis
Brief Title: Study of AROSOD-1 in Adult Participants With Amyotrophic Lateral Sclerosis (ALS)
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Company business decision
Sponsor: Arrowhead Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AROSOD1-1001; 2023-509032-26 (EudraCT Number)
Record Dates: First submitted 2023-07-08; First posted 2023-07-18 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- ARO-SOD1 (Experimental): ARO-SOD1 Injection
  Interventions: Drug: ARO-SOD1 Injection

INTERVENTIONS:
Drug: ARO-SOD1 Injection — single doses of ARO-SOD1 Injection by IT infusion

SUMMARY:
In this Phase 1 adult symptomatic patients with amyotrophic lateral sclerosis (ALS) carrying a superoxide dismutase 1 (SOD1) gene mutation thought to be causative of ALS, will receive single ascending doses of ARO-SOD1 administered by intrathecal (IT) infusion. The study is primarily intended to evaluate safety, but will also evaluate the effect of ARO-SOD1 on SOD1 cerebrospinal fluid (CSF) levels as a biomarker of pharmacodynamic (PD) effect, therefore lumbar punctures will be required at timepoints throughout the study. After each participant has completed their individual final visit, participants whose SOD1 CSF levels have recovered to a satisfactory level may rescreen and enroll into higher dose cohorts; or if unable or unwilling to rescreen may enroll into an open-label study to be added by amendment when supported by nonclinical data for multidose administration.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ALS based on source-verifiable medical record and meets the Gold Coast Criteria
* Pathogenic or likely pathogenic SOD1 mutation based on source-verifiable medical records or genetic testing during Screening
* Slow Vital Capacity (SVC) ≥ 50% of predicted value adjusted for sex, age, and height (from a sitting position) at Screening
* Body Mass Index (BMI) ≥ 18.0 kg/m2 at Screening
* Able to complete at least 6 months of follow-up
* If taking any medication or supplement to treat ALS or ALS symptoms, must be on stable dose for ≥ 4 weeks prior to Day 1 and expected to remain at that dose until final study visit and not expected to start these medications after the first dose of ARO-SOD1
* Able and willing to provide written informed consent and to comply with all study assessments
* Participants of childbearing potential must agree to use highly effective contraception in addition to a condom during the study and for at least 90 days following the end of study or last dose of study drug, whichever is later. Males must not donate sperm and females must not donate eggs during the study and for at least 90 days following the end of the study or last dose of study drug, whichever is later.

Exclusion Criteria:

* Current or anticipated need of a diaphragm pacing system (DPS) during the study
* Participants using tofersen can be enrolled only after a washout period of approximately 20 weeks from the last tofersen dose to the first planned dose of ARO-SOD1
* History of having received stem cell therapy for ALS treatment
* Any current or anticipated contraindications to lumbar puncture (LP)
* The presence of an implanted shunt for drainage of CSF or an implanted central nervous system (CNS) catheter
* Human immunodeficiency virus (HIV), seropositive for hepatitis B virus (HBV), seropositive for hepatitis C virus (HCV)
* Uncontrolled hypertension
* Severe cardiovascular disease
* History of drug abuse or alcoholism within 6 months of study enrollment
* Inability to comply with study requirements

Note: additional inclusion/exclusion criteria may apply per protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-01 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Treatment-Emergent Adverse Events (TEAEs) | From first dose of study drug through the end of study (EOS; up to 168 days)

SECONDARY OUTCOMES:
Change Over Time from Baseline in CSF SOD1 Protein Levels | Pre-dose on Day 1 (Baseline) through EOS (up to 168 days)
Change Over Time from Baseline in Plasma Levels of Neurofilament Light Chain (NfL) | Pre-dose on Day 1 (Baseline) through EOS (up to 168 days)
Pharmacokinetics (PK) of ARO-SOD1: Maximum Observed Plasma Concentration (Cmax) | Days 1, 2, 15, 29, 57, 85 and EOS (Day 168): Pre-dose, post-dose at 1, 3, 5, 7, 12 and 24 hours
PK of ARO-SOD1: Time to Reach Maximum Observed Plasma Concentration (Tmax) | Days 1, 2, 15, 29, 57, 85 and EOS (Day 168): Pre-dose, post-dose at 1, 3, 5, 7, 12 and 24 hours
PK of ARO-SOD1: Area Under the Plasma Concentration Versus Time Curve from Zero to 24 Hours (AUC0-24) | Days 1, 2, 15, 29, 57, 85 and EOS (Day 168): Pre-dose, post-dose at 1, 3, 5, 7, 12 and 24 hours
PK of ARO-SOD1: Area Under the Plasma Concentration Versus Time Curve from Zero to the Last Quantifiable Plasma Concentration (AUClast) | Days 1, 2, 15, 29, 57, 85 and EOS (Day 168): Pre-dose, post-dose at 1, 3, 5, 7, 12 and 24 hours
PK of ARO-SOD1: Area Under the Plasma Concentration Versus Time Curve from Zero to Infinity (AUCinf) | Days 1, 2, 15, 29, 57, 85 and EOS (Day 168): Pre-dose, post-dose at 1, 3, 5, 7, 12 and 24 hours
PK of ARO-SOD1: Terminal Elimination Half-Life (t1/2) | Days 1, 2, 15, 29, 57, 85 and EOS (Day 168): Pre-dose, post-dose at 1, 3, 5, 7, 12 and 24 hours
PK of ARO-SOD1: Apparent Systemic Clearance (CL/F) | Days 1, 2, 15, 29, 57, 85 and EOS (Day 168): Pre-dose, post-dose at 1, 3, 5, 7, 12 and 24 hours
PK of ARO-SOD1: Recovery of Unchanged Drug in Urine Over 0-24 Hours (Amount Excreted: Ae) | Pre-dose through 24 hours post-dose
PK of ARO-SOD1: Percentage of Administered Drug Recovered in Urine Over 0-24 Hours | Pre-dose through 24 hours post-dose
PK of ARO-SOD1: Renal Clearance (CLr) | Pre-dose through 24 hours post-dose
Change From Baseline in Total Protein in CSF | Pre-dose on Day 1 (Baseline) through EOS (up to 168 days)
Change From Baseline in Glucose in CSF | Pre-dose on Day 1 (Baseline) through EOS (up to 168 days)
Change From Baseline in Cell Count in CSF | Pre-dose on Day 1 (Baseline) through EOS (up to 168 days)

IPD SHARING:
Plan to Share IPD: No